CLINICAL TRIAL: NCT07323368
Title: Advancing Reperfusion Therapy for Ischemic Stroke (ARTS): Perfusion-guided Endovascular Intervention for Medium Vessel Occlusion Therapy (PIVOT)
Brief Title: Advancing Reperfusion Therapy for Ischemic Stroke: Perfusion-guided Endovascular Intervention for Medium Vessel Occlusion Therapy
Acronym: ARTS-PIVOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yunyun Xiong, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SQ2024QB01857
Record Dates: First submitted 2025-12-10; First posted 2026-01-07 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Stroke Ischemic; Medium Vessel Occlusions
Keywords: ischemic stroke; medium vessel occlusions; endovascular treatment; perfusion imaging
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endovascular treatment (EVT) +Best medical treatment (Experimental): The treating physician should attempt to perform EVT with the goal to restore blood flow to the affected vascular territory immediately after randomisation. EVT included thrombectomy with stent retrievers, thromboaspiration, intraarterial thrombolysis, balloon angioplasty, stenting, or a combination of these approaches at the discretion of the interventional team. All decisions regarding the performance of EVT are made by the treating physician, based on his/her own judgement, and using local standards for endovascular treatment technique and devices and/or medications used for EVT. All other treatments (especially after-care and best medical treatment) will not differ between the intervention and control group.
  Interventions: Procedure: Endovascular treatment
- Best medical treatment (BMT) (Other): Administration of BMT should be done according to routine clinical practice and current guidelines.
  Interventions: Drug: Best medical treatment (BMT)

INTERVENTIONS:
Procedure: Endovascular treatment — EVT included thrombectomy with stent retrievers, thromboaspiration, intraarterial thrombolysis, balloon angioplasty, stenting, or a combination of these approaches at the discretion of the interventional team.
  Arms: Endovascular treatment (EVT) +Best medical treatment
Drug: Best medical treatment (BMT) — Administration of BMT should be done according to routine clinical practice and current international guidelines. Administration of BMT must not be delayed by randomisation and should be done independently from participation in this trial.
  Arms: Best medical treatment (BMT)

SUMMARY:
The investigators initiated a multicenter, prospective, randomized, open label, blinded-endpoint (PROBE) controlled trial to evaluate the efficacy and safety of perfusion-guided endovascular treatment (EVT) compared to standard medical care for patients with acute ischemic stroke due to medium vessel occlusion (MeVO) within 24 hours from symptom onset.

DETAILED DESCRIPTION:
Adult acute ischemic stroke patients due to primary medium vessel occlusions (non-dominant proximal M2 or mid-distal M2/M3 segments of the middle cerebral artery, A1/A2/A3 segments of the anterior cerebral artery, and P1/P2/P3 segments of the posterior cerebral artery) confirmed by CTA/MRA and responsible for the signs and symptoms of acute ischemic stroke with baseline National Institutes of Health Stroke Scale (NIHSS) ≥8 will be enrolled in this trial. The investigators use perfusion imaging to select subjects and the enrolled patients have target mismatch profile on CTP or MRI+PWI (ischemic core volume <70mL, mismatch ratio>1.2, mismatch volume >10mL). The eligible patients will be randomly assigned to receive endovascular treatment (EVT) +best medical treatment or best medical treatment within 24 hours after the time that the patient was last known to be well (including after stroke on awakening and unwitnessed stroke). The primary outcome is the proportion of patients with an mRS score ≤ 1 at 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years old;
* Acute ischemic stroke symptom onset within 24 hours; including wake-up stroke and unwitnessed stroke, onset time refers to "last-seen normal time";
* Primary medium vessel occlusions confirmed by CTA/MRA, including non-dominant proximal M2 or mid-distal M2/M3 segments of the middle cerebral artery (MCA), A1/A2/A3 segments of the anterior cerebral artery (ACA), and P1/P2/P3 segments of the posterior cerebral artery (PCA) and responsible for the signs and symptoms of acute ischemic stroke;
* Pre-stroke modified Rankin scale (mRS) score ≤1;
* Baseline National Institutes of Health Stroke Scale (NIHSS) ≥8;
* Neuroimaging criteria: Target mismatch profile on CT perfusion or MRI+MR perfusion (ischemic core volume <70 mL, mismatch rate >1.2, mismatch volume >10 mL);
* Written informed consent from patients or their legally authorized representatives.

Exclusion Criteria:

* Any evidence of intracranial hemorrhage on qualifying imaging;
* Known (serious) sensitivity to radiographic contrast agents, nickel, titanium metals or their alloys and unable to complete CTP/PWI;
* Known history of arterial tortuosity, pre-existing stent, other arterial disease and/or known disease at the arterial access site that would prevent the device from reaching the target vessel and/or preclude safe recovery after EVT;
* Radiological confirmed evidence of mass effect or intracranial tumour (except small meningioma);
* Clinical diagnosis of cerebral vasculitis;
* Evidence of vessel recanalization prior to randomisation;
* Severe comorbidities, which will likely prevent improvement or follow-up;
* Any terminal illness such that the patient would not be expected to survive more than 1 year;
* Hypodensity in >1/3 MCA territory on non-contrast CT or significant hypodensity outside the current perfusion lesion suggesting distal clot migration (secondary MeVO);
* Multiple arterial occlusion;
* Pregnant women, nursing mothers, or reluctance to use effective contraceptive measures during the period of the trial;
* Unlikely to adhere to the trial protocol or follow-up;
* Participation in other interventional clinical trials within the previous 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 568 (Estimated)
Dates: Start 2026-02-08 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients who have a score of 0 or 1 on the modified Rankin Scale (mRS) at 90 days | 90 days
  The proportion of patients with an mRS score ≤ 1 at 90 days. The mRS score is a seven-point ordered categorical scale from 0 to 6 for functional neurological outcome, with 0 indicating no neurological symptoms and 6 indicating death.

SECONDARY OUTCOMES:
Ordinal distribution of modified Rankin Scale (mRS) at 90 days | 90 days
  Ordinal distribution of mRS at 90 days (shift analysis). The mRS score is a seven-point ordered categorical scale from 0 to 6 for functional neurological outcome, with 0 indicating no neurological symptoms and 6 indicating death.
The proportion of patients with an modified Rankin Scale (mRS) score of 0-2 at 90 days | 90 days
  The proportion of patients with an mRS score of 0-2 at 90 days. The mRS score is a seven-point ordered categorical scale from 0 to 6 for functional neurological outcome, with 0 indicating no neurological symptoms and 6 indicating death.
The rate of early neurological improvement at 24 hours | 24 hours
  The rate of early neurological improvement at 24 hours after randomization (defined as a National Institute of Health Stroke Scale [NIHSS] score ≤1 or ≥4 points compared with the baseline)
The proportion of patients with an modified Rankin Scale (mRS) score of 5-6 at 90 days | 90 days
  The proportion of patients with an mRS score of 0-2 at 90 days. The mRS score is a seven-point ordered categorical scale from 0 to 6 for functional neurological outcome, with 0 indicating no neurological symptoms and 6 indicating death.
The median value of EuroQol 5-Dimension (EQ-5D) index | 90 days and 1 year
  EuroQol 5-Dimension (EQ-5D) index at 90 days and 1 year. The EuroQol Group 5-Dimension Self-Report Questionnaire (EQ-5D) is a standardized instrument for the measurement of health status. The domains mobility, self-care, everyday activity, pain or physical discomfort, and fear or depression are assessed on a five-point scale, with 1 indicating no problem in this domain and 3 indicating extreme problems. The visual analogue scale ranges from 0 to 100, with 0 indicating the worst health imaginable and 100 the best health imaginable.
Ordinal distribution of modified Rankin Scale (mRS) at 1 year | 1 year
  Ordinal distribution of modified Rankin Scale (mRS) at 90 days. The mRS score is a seven-point ordered categorical scale from 0 to 6 for functional neurological outcome, with 0 indicating no neurological symptoms and 6 indicating death.
The proportion of symptomatic intracranial hemorrhage | 24 hours
  Symptomatic intracranial hemorrhage within 24 hours (as defined by Heidelberg criteria)
The proportion of all-cause mortality | 90 days and 1 year
  All-cause mortality at 90 days and 1 year
The proportion of systematic bleeding | 90 days
  Moderate or severe systemic bleeding is defined according to the criteria established in the Global Utilization of Streptokinase and Tissue Plasminogen Activator for Occluded Coronary Arteries (GUSTO) trial
The proportion of serious adverse events (SAEs) | 90 days
  serious adverse events within 90 days

OTHER OUTCOMES:
The proportion of successful recanalization | immediately after the intervention
  The proportion of successful recanalization(eTICI 2b50-3) following EVT
The proportion of improvement on reperfusion at 24 hours after randomization | 24 hours
  Improvement on reperfusion is defined as >90% reduction in Tmax > 6s lesion volume
The proportion of complete recanalization at 24 hours after randomization | 24 hours
  Complete recanalization is defined as an Arterial Occlusion Lesion scale [AOL] score of 3 (scale range, 0 [no recanalization] to 3 [complete recanalization]).

CONTACTS AND LOCATIONS:
Overall Officials: Yunyun Xiong, professor, Principal Investigator — Beijing Tiantan Hospital
Locations (6):
- China (6):
  - Beijing tiantan hospital, Beijing, Beijing Municipality
  - Beijing Daxing District People's Hospital, Beijing, Beijing Municipality
  - Xingtang County People's Hospital, Longzhou, Hebei
  - Luoyang Yiluo Hospital, Luoyang, Henan
  - People's Hospital of Queshan, Panlong, Henan
  - Changle People's Hospital, Changle, Shandong

IPD SHARING:
Plan to Share IPD: Undecided